CLINICAL TRIAL: NCT07145502
Title: Monitoring of Outcomes of Cellular and Exosome-based Therapies in Autoinflammatory and Post-infectious Neuroinflammatory Syndromes
Status: Active, not recruiting | Type: Observational
Sponsor: Biocells Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Bio120001
Record Dates: First submitted 2025-06-08; First posted 2025-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Encephalitis; Early-stage Panencephalitis; Neuroinflammatory Demyelination
Keywords: Autoimmune encephalitis; Early-stage panencephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- B1: * Age 6-70
  * Diagnosis of one of the eligible syndromes by neurologist or immunologist
  * Unresponsive or partially responsive to conventional therapy
  * Informed consent provided
  Interventions: Biological: Allogeneic MSC infusions (IV)

INTERVENTIONS:
Biological: Allogeneic MSC infusions (IV) — Optional T-reg therapy (experimental/compassionate-use basis)
  Other Names: MSC-derived exosomes (IV or intranasal); Supportive immunomodulatory agents

SUMMARY:
This is a prospective, non-randomized, observational registry study evaluating the clinical outcomes of patients with autoimmune or post-infectious neuroinflammatory syndromes receiving stem cell-derived biologics (including mesenchymal stem cells and exosomes) at Biocells Medical clinics. The study aims to track improvements in neurological function, inflammatory biomarkers, and patient-reported quality of life following individualized regenerative interventions.

ELIGIBILITY:
Inclusion Criteria:

* • Age 6-70

  * Diagnosis of one of the eligible syndromes by neurologist or immunologist
  * Unresponsive or partially responsive to conventional therapy
  * Informed consent provided

Exclusion Criteria:

* • Active malignancy

  * Severe systemic infection
  * Contraindications to IV biologics

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include pediatric, adult, and older adult patients aged 6 to 70 years who present with clinically confirmed or strongly suspected neuroinflammatory conditions of autoimmune or post-infectious origin. These include but are not limited to autoimmune encephalitis, post-viral encephalopathies (e.g., following measles, CMV, EBV, SARS-CoV-2), early-stage panencephalitis, and chronic neuroimmune syndromes such as ME/CFS and long COVID with CNS involvement.
  Patients are eligible for inclusion if they have a persistent neuroinflammatory or neurocognitive condition that has not responded adequately to standard therapies or has relapsed. Diagnostic confirmation may include MRI findings, CSF analysis, neuropsychological testing, and immunological profiling (e.g., autoantibodies, cytokines).
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2027-09-19 (Estimated)

PRIMARY OUTCOMES:
Change in neurological symptom severity | from enrollment to the end of treatment at 8 weeks
  Change in neurological symptom severity as measured by the National Institutes of Health Stroke Scale (NIHSS; range 0-42, higher scores indicate greater severity)

SECONDARY OUTCOMES:
Change in serum cytokine levels | From the enrolment till the end of the treatment (8 weeks)
  IL-6, TNF-α, pg/mL
Change in patient-reported quality of life | From the enrolment to the end of the treatment (8 weeks)
  EQ-5D (range: 5-25, lower scores indicate better health-related quality of life)
Change in patient-reported quality of life | From the enrolment till the end of the treatment (8 weeks)
  SF-36 (range: 0-100, higher scores indicate better health-related quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Biocells Medical, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided